CLINICAL TRIAL: NCT07096401
Title: The Efficacy of Aligner Therapy Versus Anterior Bite Turbos and Reverse Curve of Spee Archwires for Correction of Deep Bite Cases: A Cone-beam Computed Tomography Study
Brief Title: Efficacy of Aligners vs ABT and RCOS for Deep Bite Correction: CBCT Study
Acronym: DB-CBCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hisham Alaa Eldien Elsayed Ahmed, The efficacy of aligner therapy versus two different methods for correction of deep bite cases. cone-beam computed tomography study, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AU-Ortho-DB-2025
Record Dates: First submitted 2025-07-16; First posted 2025-07-31 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Deep Bite Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RCOS Archwire Group (Experimental): Patients treated with reverse curve of Spee archwire (0.016 × 0.022 NiTi) to correct deep bite via posterior extrusion and anterior intrusion.
  Interventions: Device: Reverse Curve of Spee Archwire
- Anterior Bite Turbos Group (Experimental): Patients treated with anterior bite turbos bonded to the palatal surface of upper central incisors to correct deep bite.
  Interventions: Device: Anterior Bite Turbos
- Clear Aligners Group (Experimental)
  Interventions: Device: Clear Aligners

INTERVENTIONS:
Device: Reverse Curve of Spee Archwire — Orthodontic treatment using a 0.016 × 0.022 NiTi reverse curve of Spee archwire to correct deep bite through posterior extrusion and anterior intrusion.
  Arms: RCOS Archwire Group
Device: Anterior Bite Turbos — Orthodontic treatment using anterior bite turbos bonded to the palatal surfaces of the upper central incisors to promote posterior extrusion and correct deep bite.
  Arms: Anterior Bite Turbos Group
Device: Clear Aligners — Orthodontic treatment using clear aligner therapy designed for anterior intrusion and leveling of the curve of Spee to correct deep bite.
  Arms: Clear Aligners Group

SUMMARY:
This prospective clinical trial aims to evaluate the efficacy of clear aligner therapy compared to two different treatment modalities - anterior bite turbos and reverse curve of Spee (RCOS) archwires - for the correction of dental deep bite cases. Deep bite malocclusion is characterized by excessive vertical overlap of the anterior teeth and often requires intrusion of anterior teeth and leveling of the curve of Spee.

In this study, 27 patients aged 16-30 years with an overbite ≥5 mm and no significant skeletal discrepancies will be randomly assigned into three equal groups: Group 1 (RCOS archwire), Group 2 (anterior bite turbos), and Group 3 (clear aligners).

Cone-beam computed tomography (CBCT) will be used to assess changes in overbite and alveolar bone height and thickness before and after treatment. The primary outcome is the efficacy of overbite correction, and the secondary outcome is the assessment of alveolar bone remodeling.

The study will be conducted at the Department of Orthodontics, Faculty of Dental Medicine, Al-Azhar University (Assiut Branch), and has been approved by the institutional ethical committee.

ELIGIBILITY:
Inclusion Criteria:

- Age between 16 and 30 years.

Overbite of 5 mm or more.

Full permanent dentition (excluding third molars).

Good oral hygiene.

No previous orthodontic or orthognathic treatment.

Exclusion Criteria:

* Severe skeletal Class II or III requiring surgery.

Overjet greater than 6 mm.

Craniofacial anomalies.

Systemic diseases.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 27 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in overbite | Baseline and 6 months after treatment start
  Mean change in overbite (in mm) measured using CBCT imaging